CLINICAL TRIAL: NCT05842473
Title: Long-term Effect of Transcranial Magnetic Stimulation in Primary Progressive Aphasia
Brief Title: Long-term Effect of TMS in Primary Progressive Aphasia
Acronym: RECONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jordi A Matias-Guiu, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21/731-EC_P
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Primary Progressive Aphasia; Frontotemporal Dementia; Alzheimer Disease
Keywords: brain stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Alzheimer Disease | interventions — Transcranial Magnetic Stimulation; Language Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMS active + language therapy (Active Comparator): TMS (active) using theta burst protocol over the left dorsolateral prefrontal cortex. Daily sessions for two weeks followed by one session per week during 6 months. Each TMS session is followed by language training.
  Interventions: Device: Transcranial Magnetic Stimulation (active); Behavioral: Language therapy
- TMS sham + language therapy (Sham Comparator): TMS (sham) using theta burst protocol over the left dorsolateral prefrontal cortex. Daily sessions for two weeks followed by one session per week during 6 months. Each TMS session is followed by language training.
  Interventions: Behavioral: Language therapy; Device: Transcranial Magnetic Stimulation (sham)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (active) — Theta-burst transcranial magnetic stimulation (active) delivered over the left dorsolateral prefrontal cortex. Daily sessions for two weeks followed by 1 session per week.
  Arms: TMS active + language therapy
Behavioral: Language therapy — Language therapy immediately after each TMS session. Daily sessions for two weeks followed by 1 session per week.
Device: Transcranial Magnetic Stimulation (sham) — Theta-burst transcranial magnetic stimulation (sham) delivered over the left dorsolateral prefrontal cortex. Daily sessions for two weeks followed by 1 session per week.
  Arms: TMS sham + language therapy

SUMMARY:
There are very few treatments for neurodegenerative disorders, and the efficacy of these treatments is generally modest. Recent studies have shown a short-term positive effect of non-invasive neuromodulation techniques such as transcranial magnetic stimulation (TMS) in primary progressive aphasia (PPA). PPA is a clinical syndrome associated with Alzheimer's disease and Frontotemporal degeneration. The aim of this study is to compare the effect of TMS and language therapy versus language therapy and sham TMS in patients with PPA during 6 months. A prospective, randomized, controlled, double-blind and parallel clinical trial will be conducted. The changes in brain metabolism using FDG-PET, language, neuropsychiatric symptoms, and daily-living activities will be assessed. Connectivity changes using electroencephalography will also be examined. In addition, a subgroup of patients will be assessed with multimodal MRI (structural and functional), and blood biomarkers. As a result of this project, valuable information about the long-term efficacy of non-invasive brain stimulation in PPA will be obtained, as well as the mechanisms of the therapy and clinical and neuroimaging factors associated with therapy response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA (Gorno-Tempini et al. 2011 criteria supported by neuroimaging)
* CDR
* Language is the most prominent symptom

Exclusion Criteria:

* Clinical Dementia Rating scale > 1
* History of epilepsy or epileptiform activity in EEG
* Another disorder causing aphasia
* Any contraindication for TMS
* Pregnancy
* Medical disorder with a life expectancy of less than one year
* Malignancy in the last two years
* Alcohol or drug abuse
* Major psychiatric disorder
* Inability to communicate (mutism)
* Use of anticonvulsants, benzodiazepines, donepezil/galantamine/rivastigmine, memantine, antidepressants and neuroleptics is permitted if they are at stable doses in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Brain Metabolism | 0 and 6 months
  Changes in FDG-PET imaging (Standard Uptake Value ratio)

SECONDARY OUTCOMES:
Spontaneous language | 0, 3 and 6 months
  Changes in Words per minute
Language assessment (Mini-Linguistic State Examination) | 0, 3 and 6 months
  Changes in Mini-Linguistic State Examination test
Language assessment (trained words) | 0, 3 and 6 months
  Changes in trained words accuracy (number of words)
Daily-living activities | 0, 3 and 6 months
  Changes in Interview for Deterioration in Daily living in Dementia Scale
Neuropsychiatric symptoms | 0, 3 and 6 months
  Changes in Neuropsychiatric Inventory scale

CONTACTS AND LOCATIONS:
Overall Officials: Jordi A Matias-Guiu, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clínico San Carlos., Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fernandez-Romero L, Cabrera-Martin MN, Delgado-Alonso C, Suarez-Coalla P, Grasso SM, Portoles A, Perez-Macias N, Carreras MT, Diez-Cirarda M, Gil-Moreno MJ, Olazaran J, Vieira A, Oliver-Mas S, Gomez-Pinedo U, Matias-Guiu J, Matias-Guiu JA. Long-Term Therapy With Transcranial Magnetic Stimulation in Primary Progressive Aphasia: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526129. doi: 10.1001/jamanetworkopen.2025.26129. PMID 40788648